CLINICAL TRIAL: NCT04243408
Title: Treatment of Children With Cerebral Palsy With Autologous Umbilical Cord Blood, a Pilot Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Omer Bar-Yosef, M.D.-Ph.D. Peadiatric Neurology and Child Development. Deputy Director The Edmond and Lily Safra Children's Hospital, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHEBA-18-5102-OBY-CTIL
Record Dates: First submitted 2020-01-15; First posted 2020-01-28 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy, autologous umbilical cord blood
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: This study is a phase II, prospective, double blind, placebo-control study of the efficacy of autologous umbilical cord blood infusion.
  The study population will consist of 72 children ages 2 months to 12 years with cerebral palsy. The population will be randomly assigned to 2 groups, the study group be treated by cord blood in the beginning of the study and the control group by placebo product.
  The study population will be stratified to reduce variance 3 groups by age: 2-12 months / 1-6 years / 6-12 years The study will consist of 4 stages Stage 1: initial assessment by physiotherapist and occupational therapist / treatment by cord blood or placebo / blood work before and after treatment Stage 2: at stage 1 + 3 months assessment by physiotherapist and occupational therapist Stage 3: at stage 1 + 6 months assessment by physiotherapist and occupational therapist
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization will be done by external source and the assignment will disclosed to cord bank bank only. They will produce either a cord blood or placebo unit which will be completely covered. Each unit will have its own index number that will be documented by the research coordinator. Neither the researcher or the family will know the nature of the unit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group 1 (Experimental)
  Interventions: Other: Autologous umbilical cord blood transfusion
- group 2 (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Other: Autologous umbilical cord blood transfusion — single dose of an autologous umbilical cord blood transfusion
  Arms: group 1
Other: placebo — The placebo product will consist of the standard ingredients of the acellular content of the UCB unit. It will consist of 20 ml Dextran (Plander 40.000 - 50g/500ml, solution for infusion) and 20 ml of human Albumin 5% (solution for infusion). The volume of placebo product will be 40 ml
  Arms: group 2

SUMMARY:
This study is a phase II, prospective, double blind, placebo-controlled study of the efficacy of autologous umbilical cord blood infusion.

The study population will consist of 72 children ages 2 months to 12 years with cerebral palsy. The population will be randomly assigned to 2 groups, 36 children in each group. The study group be treated by cord blood in the beginning of the study and the control group by placebo product. The study population will be stratified to reduce variance 3 groups by age: 2-12 months / 1-6 years / 6-12 years The study will consist of 4 stages Stage 1: initial assessment by physiotherapist and occupational therapist / treatment by cord blood or placebo / blood work before and after treatment Stage 2: at stage 1 + 3 months assessment by physiotherapist and occupational therapist Stage 3: at stage 1 + 6 months assessment by physiotherapist and occupational therapist / cross-over treatment by cord blood or placebo / blood work before and after treatment Stage 4: at stage 1 + 12 months assessment by physiotherapist and occupational therapist The primary outcome is improvement motor skills six months after treatment at stage 3

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 2 month and ≤ 12 years.
* Performance status for children older than 2 months and younger than 12 months including all the following (Gross Motor Function Classification Score is less indicative before 12 months):

  * Abnormal General Movements (in infants 2-6 months)
  * Abnormal Hammersmith Infant Neurological Examination
* Performance status for children older than 12 months

  * Bilateral spastic cerebral palsy (diplegia or quadraplegia): Gross Motor Function Classification Score levels I - IV
  * Spastic hemiplegia: Gross Motor Function Classification Score levels I - IV. A subject classified as GMFCS level I with significant upper extremity impairment will be eligible if the affected upper extremity is used as an assist only.
  * Bilateral hypotonic cerebral palsy (diplegia or quadraplegia): Gross Motor Function Classification Score levels I - IV.
* An abnormal brain MRI suggestive of an acquired etiology (and not genetic etiology or brain malformation).
* 4. Autologous umbilical cord blood available at a private or public cord blood bank with a minimum total nucleated cell dose of ≥ 2 x 10e7 cells/kilogram.
* 5. Parental consent.

Exclusion Criteria:

* Autism and autistic spectrum disorders without motor disability.
* Hypsarrhythmia.
* Intractable seizures causing epileptic encephalopathy.
* Evidence of a progressive neurologic disease.
* Known HIV or uncontrolled bacterial, fungal, or viral infections.
* Impaired renal or liver function as determined by serum creatinine >1.5mg/dL and/or total bilirubin >1.3mg/dL.
* Head circumference >3 standard deviations below the mean for age.
* Known genetic disease or phenotypic evidence of a genetic disease on physical examination.
* Requires ventilatory support, including home ventilator
* Surgical procedure or botulinum toxin injection from 6 months prior to the study and during the time of the study
* Patient's medical condition does not permit safe travel.
* Previously received any form of cellular therapy.

  * Autologous umbilical cord blood unit has any of the following:
  * Total nuclear cell dose < 2 x 10e7 cells/kilogram
  * Positive maternal infectious disease markers (except CMV)
  * Evidence of infectious contamination of the cord blood unit
* Lack of a test sample to confirm identity
* Evidence of a genetic disease
* Unable to obtain parental consent.

Ages: 2 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2020-07-08 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Motor developmental improvement | 6 months
  Gross Motor Function Measurement - 66 (GMFM-66). All score are normalized with mean 100 and STD of 15. High score is better than low score .
Motor developmental improvement | 6 months
  Peabody developmental motor scales-second edition (PDMS-2). All score are normalized with mean 100 and STD 10. High score is better
Functional assessment | 6 months
  Pediatric Evaluation of Disability Evaluation . Score 0-100 higher score better functionality Pediatric Evaluation of Disability Inventory-Computer Adaptive Test (PEDI-CAT)

SECONDARY OUTCOMES:
Functional assessment | 6 months
  Adaptive Behavior Assessment System, Third Edition (ABAS-3). All score are normalized with mean 100 and STD of 10. High score is better than low score .
Functional assessment | 6 months
  Vineland Adaptive Behavior Scales-Second Edition (VINELAND-II). All score are normalized with mean 100 and STD of 15. High score is better than low score .

CONTACTS AND LOCATIONS:
Overall Officials: Omer Bar-Yosef, MD.PHD, Study Director — Sheba Medical Center
Locations (1):
- Chaim Seba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Yes
data set of the baseline of the children, the quantity of cord blood transfusion they received and the clinical followup information.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: within 2 years from the end of data collection

REFERENCES:
- [Background] Bax M, Goldstein M, Rosenbaum P, Leviton A, Paneth N, Dan B, Jacobsson B, Damiano D; Executive Committee for the Definition of Cerebral Palsy. Proposed definition and classification of cerebral palsy, April 2005. Dev Med Child Neurol. 2005 Aug;47(8):571-6. doi: 10.1017/s001216220500112x. PMID 16108461
- [Background] Colver A, Fairhurst C, Pharoah PO. Cerebral palsy. Lancet. 2014 Apr 5;383(9924):1240-9. doi: 10.1016/S0140-6736(13)61835-8. Epub 2013 Nov 20. PMID 24268104
- [Background] Clark SL, Hankins GD. Temporal and demographic trends in cerebral palsy--fact and fiction. Am J Obstet Gynecol. 2003 Mar;188(3):628-33. doi: 10.1067/mob.2003.204. PMID 12634632